CLINICAL TRIAL: NCT06271265
Title: A Multicenter, Open-label, Randomized, Bupivacaine-Controlled Study to Evaluate the Pharmacokinetics and Safety of EXPAREL for Postoperative Analgesia in Subjects Aged 0 to Less Than 6 Years Undergoing Cardiac Surgery
Brief Title: Study to Evaluate the Pharmacokinetics and Safety of EXPAREL for Postoperative Analgesia in Subjects Undergoing Cardiac Surgery
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-125
Record Dates: First submitted 2024-01-18; First posted 2024-02-21 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain
Keywords: Analgesia; Cardiac Surgery; Pediatric
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EXPAREL (Experimental): A total of approximately 24 subjects (8 subjects per Part) will be enrolled. Subjects in this arm will receive EXPAREL
  Interventions: Drug: EXPAREL
- bupivacaine (Active Comparator): A total of approximately 24 subjects (8 subjects per Part) will be enrolled. Subjects in this arm will receive bupivacaine
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: EXPAREL — A single dose of EXPAREL Injectable Product via LIA
  Arms: EXPAREL
Drug: bupivacaine — A single dose of 0.25% bupivacaine via LIA
  Arms: bupivacaine

SUMMARY:
This Phase 1, multicenter, open-label, randomized, bupivacaine-controlled study is designed to evaluate the pharmacokinetics (PK) and safety of EXPAREL vs. bupivacaine HCl for postsurgical analgesia in pediatric subjects aged 0 to less than 6 years of age undergoing cardiac surgery, utilizing local infiltration analgesia (LIA).

DETAILED DESCRIPTION:
This study will be conducted in 3 Parts (Part 1, Part 2, and Part 3) and a total of approximately 48 male and female subjects will be enrolled.

Part 1 will enroll approximately 16 subjects, aged 2 to less than 6 years to obtain information on PK and safety. Subjects will be randomized 1:1 (8 EXPAREL subjects and 8 bupivacaine HCl subjects) to receive either a single dose of EXPAREL 4 mg/kg (not to exceed a maximum total dose of 266 mg) or 0.25% bupivacaine HCl 2 mg/kg (not to exceed a maximum total dose of 175 mg) using LIA. The overall PK and safety profiles from Part 1 will be completed, analyzed, and reviewed to establish an appropriate study drug dose for Part 2.

Subject enrollment for Part 2 will commence upon complete enrollment of Part 1, establishment of an appropriate study drug dose from the PK, and safety analysis of Part 1 and Data Safety Monitoring Board (DSMB) recommendations to proceed to Part 2. Part 2 will enroll approximately 16 subjects, aged 6 months to less than 2 years to obtain information on PK and safety. Subjects will be randomized 1:1 (8 EXPAREL subjects and 8 bupivacaine HCl subjects) to receive either a single dose of EXPAREL or 0.25% bupivacaine HCl using LIA. The overall PK and safety profiles from Part 2 will be completed, analyzed, and reviewed to establish an appropriate study drug dose for Part 3.

Subject enrollment for Part 3 will commence upon complete enrollment of Part 2, establishment of an appropriate study drug dose from the PK and safety analysis of Part 2, and DSMB recommendations to proceed to Part 3.

Part 3 will enroll approximately 16 subjects aged 0 to less than 6 months to obtain information on PK and safety. Subjects will be randomized 1:1 (8 EXPAREL subjects and 8 bupivacaine HCL subjects) to receive either a single dose of EXPAREL or 0.25% bupivacaine HCl using LIA.

ELIGIBILITY:
Inclusion Criteria:

All of the following inclusion criteria must be met for eligibility:

1. Pediatric participants with congenital heart defects planned to undergo cardiac surgery with cardiopulmonary bypass
2. Male or female participants from 0 to less than 6 years of age on the day of surgery: 2 years to less than 6 years of age for Part 1; 6 months to less than 2 years of age for Part 2; 0 to less than 6 months of age for Part 3
3. American Society of Anesthesiologists (ASA) Classes 1 through 4.
4. Parent/guardian is able to speak, read, and understand the language of the ICF and provide informed consent for the participant.
5. Parent/guardian is able to adhere to the study visit schedule and complete all study assessments for the participant.

Exclusion Criteria:

Exclusion Criteria:

A participant will not be eligible for the study if any of the following exclusion criteria are met:

1. History of hypersensitivity or idiosyncratic reactions or contradictions to EXPAREL, bupivacaine HCl, or other amide-type local anesthetics or to opioid medications
2. Administration of EXPAREL or bupivacaine HCl within 30 days prior to IP administration
3. Administration of an IP within 30 days or 5 elimination half-lives of such IP, whichever is longer, prior to IP administration, or planned administration of another IP or procedure during participation in this study
4. History of preterm birth (before 35 weeks of pregnancy)
5. History of coagulopathies or immunodeficiency disorders
6. Disease or condition that, in the opinion of the Investigator, indicates an increased vulnerability to IPs and/or procedures
7. Recent or potential exposure to COVID-19
8. Cardiac surgery has been canceled and cannot be rescheduled within 30 days of signing the ICF because of any reason.
9. Necessity in delayed wound closure
10. Informed consent withdrawn before randomization

Ages: 0 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The following model-predicted PK endpoint will be determined: | through 72 hours
  • Area under the plasma concentration-versus-time curve (AUClast and AUC0-inf)
The following model-predicted PK endpoint will be determined: | through 72 hours
  • Maximum observed plasma concentration (Cmax)
The following model-predicted PK endpoint will be determined: | through 72 hours
  • Time of maximum observed plasma concentration (Tmax)
The following model-predicted PK endpoint will be determined: | through 72 hours
  • The apparent terminal elimination half-life (t1/2)
The following model-predicted PK endpoint will be determined: | through 72 hours
  • Apparent clearance (CL)
The following model-predicted PK endpoint will be determined: | through 72 hours
  • Apparent volume of distribution (Vd)

SECONDARY OUTCOMES:
Vitals change from Baseline: | up to 4 postoperative days
  temperature
Vitals change from Baseline: | up to 4 postoperative days
  heart rate
Vitals change from Baseline: | up to 4 postoperative days
  respiratory rate
Vitals change from Baseline: | up to 4 postoperative days
  oxygen saturation
Vitals change from Baseline: | up to 4 postoperative days
  blood pressure
Incidence of treatment-emergent adverse events (TEAEs) | 14 ± 3 days
Incidence of adverse events of special interest (AESIs) | 14 ± 3 days
Incidence of serious adverse events (SAEs) | 14 ± 3 days

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Indiana University Health, Riley Hospital For Children, Indianapolis, Indiana
  - St. Louis Children's Hospital (SLCH), St Louis, Missouri
  - Duke University Health System, Durham, North Carolina
  - University of Oklahoma (OU) - Medical Center - The Children's Hospital, Oklahoma City, Oklahoma
  - The University of Texas Health Science Center at Houston (UTHSC-H) - McGovern Medical School, Houston, Texas